CLINICAL TRIAL: NCT03039218
Title: A Randomized, Double-Blind, Placebo-Controlled, Open-Label Extension Clinical Trial of the Dornier Aries 2 Extracorporeal Shock Wave Device for the Treatment of Mild Erectile Dysfunction (ED)
Brief Title: Dornier Aries 2 Extracorporeal Shock Wave Device for the Treatment of Mild Erectile Dysfunction (ED)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Commercial decision
Sponsor: Dornier MedTech Systems (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G140216 S004
Record Dates: First submitted 2017-01-26; First posted 2017-02-01 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Erectile Dysfunction
Keywords: erectile dysfunction; shockwave; Dornier
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Intervention Model Description: A total of 100 subjects will be randomized to either the Active or Sham/Placebo group. Following completion of the 3 month follow-up visit, subjects will be unblinded. Subjects who received the Placebo/Sham treatment will be offered treatment using the Active device applicator.
Who Masked: Participant, Investigator
Masking Description: Study subjects will be randomized in a 2:1 ratio to either active treatment or the control. The investigator and his staff do not know which applicator is the sham/placebo control and which are the active applicators. For the active treatment, a regular EMSE shockwave applicator will be used. The treatment group is further split into two equal groups, with both groups receiving the identical active treatment. In order to preserve the blinding of the investigator, the treatment devices are provided with two applicators (one for each of the active treatment groups), which while identical in function, differ slightly in appearance.
  For the sham treatment, a placebo applicator, including an absorber without emitting shockwaves, will be used. However, all three applicators (two to use with the active device and one with the sham) are going to produce exactly the typical shock wave sound with equivalent noise to reduce or eliminate bias from the investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active (Active Comparator): Subjects assigned to this group will receive Active treatments using the Dornier Aries 2.
  Interventions: Device: Dornier Aries 2
- Placebo / Sham (Placebo Comparator): Subjects assigned to this group will receive placebo / sham (no active treatment).
  Interventions: Device: Placebo / Sham

INTERVENTIONS:
Device: Dornier Aries 2 — Extracorporeal Shock Wave Device for treatment of mild erectile dysfunction
  Arms: Active
Device: Placebo / Sham — Inactive (placebo/sham) Extracorporeal Shock Wave Device for treatment of mild erectile dysfunction
  Arms: Placebo / Sham

SUMMARY:
This protocol allows for treatment of 100 men in two groups (placebo and active treatment) of 22-70 years of age with mild (IIEF EF of 17 to 25 at baseline) vasculogenic erectile dysfunction of at least 6 months duration with low intensity extracorporeal shock wave therapy utilizing the Dornier Aries 2 device.

DETAILED DESCRIPTION:
This trial is a prospective, randomized, placebo-controlled, double-blind pivotal study, with an open-label extension. The study will include 4 sites and multiple investigators. A total of 100 men with at least a 6-month history of ED and who have responded to PDE5 inhibitors will be enrolled. The trial comprises two arms to achieve equal characteristics, where patients are randomly assigned to active treatment or sham treatment.

All patients on active treatment will receive LI-ESWT treatment using the Dornier Aries 2. Patients assigned to the placebo group will receive the Dornier Aries 2 treatment using a sham applicator. The time between two treatments is 6-7 days to allow for angiogenesis and perfusion improvements to occur. The subjects' duration of participation will be a total of 34 weeks Subjects will also be asked to maintain their current level of sexual activity while participating in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate.
2. Age 22-70 years.
3. Presence of Vasculogenic Erectile Dysfunction for at least 6 months.
4. Having some response to a PDE5i. Last PDE5i use must be within 30 days of Screening Visit.
5. IIEF-EF score ≥17 up to ≤30 while taking PDE5i.
6. IIEF-EF score ≥17 up to ≤25 after wash out of PDE5i.
7. In a stable heterosexual relationship of more than three months duration.
8. Sexually active and agree to suspend all ED therapy for duration of study.
9. Agree to maintain their normal sexual habits.

Exclusion Criteria:

1. Radical prostatectomy.
2. Previous radiation therapy to pelvis.
3. Previous stem cell or platelet rich plasma therapy.
4. Previous pelvic surgeries that in the judgment of the investigator could impact on erectile function such as radical prostatectomy, radical cystectomy, Peyronie's disease surgery, penile lengthening or penile cancer surgery.
5. Untreated Hypogonadism as demonstrated by abnormal testosterone levels lower than 300 ng/dL.
6. Hormone usage, other than testosterone, clomiphene or thyroid medication.
7. Use of cocaine, cannabinoids, opiates, barbiturates, amphetamines, or benzodiazepine as demonstrated in the drug screen.
8. Psychogenic ED.
9. Peyronie's Disease or penile curvature that negatively influences sexual activity.
10. Current anticoagulation therapy or significant hematological conditions as demonstrated in abnormal values in the complete blood count.
11. Liver disease as demonstrated by abnormal chemistry panel or coagulation values in the prothrombin time (PT) along with its derived measures of prothrombin ratio (PR) blood tests.
12. Abnormal serum testosterone level defined as a value lower than 300 ng/dL or greater than 1197 ng/dL.
13. Patients with cardiac or non-cardiac electrical devices implanted.
14. Anatomical or neurological abnormalities in the treatment area.
15. Diabetes Mellitus with severe polyneuropathy.
16. Patients with generalized polyneuropathy irrespective of cause.
17. Refusal to suspend ED therapy for duration of study.
18. Men deemed not healthy enough to participate in sexual activity.
19. IIEF-EF score of 0-16 or higher than 25 at baseline assessment following "washout" period.
20. Average EHS ≤ 2 at baseline assessment following "washout".
21. Any condition or behavior that indicates to the Principal Investigator that the subject is unlikely to be compliant with study procedures and visits.
22. Any health history or laboratory result that indicates to the Principal Investigator that the subject has a significant medical condition and should not participate in the study.
23. Known allergy to ultrasound gel.

Ages: 22 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study is for males with erectile dysfunction
Enrollment: 54 (Actual)
Dates: Start 2017-02-07 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
International Inventory of Erectile Function ("IIEF") | primary outcome at 3 month follow-up visit
  validated, multi-dimensional, self-administered investigation that has been found useful in the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials

OTHER OUTCOMES:
Erectile Hardness Score | Proportion of patients with an EHS=4 at the 3 month follow-up visit
  tool to evaluate erectile dysfunction (ED) - a man's inability to get or maintain an erection firm enough for sex.
Global Assessment Questionnaire ("GAQ"). | The proportion of subjects that answer the GAQ positively through the 3 month follow-up visit
  2 question questionnaire that assesses improvement in symptoms following treatment

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Goldstein, Principal Investigator — San Diego Sexual Medicine
Locations (4):
- United States (4):
  - San Diego Sexual Medicine, San Diego, California
  - Adult Pediatric Urology & Urogynecology, Omaha, Nebraska
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Manhattan Medical Research, New York, New York

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared with other researchers.

REFERENCES:
- [Result] Clavijo RI, Kohn TP, Kohn JR, Ramasamy R. Effects of Low-Intensity Extracorporeal Shockwave Therapy on Erectile Dysfunction: A Systematic Review and Meta-Analysis. J Sex Med. 2017 Jan;14(1):27-35. doi: 10.1016/j.jsxm.2016.11.001. Epub 2016 Dec 13. PMID 27986492
- [Result] Angulo JC, Arance I, de Las Heras MM, Meilan E, Esquinas C, Andres EM. Efficacy of low-intensity shock wave therapy for erectile dysfunction: A systematic review and meta-analysis. Actas Urol Esp. 2017 Oct;41(8):479-490. doi: 10.1016/j.acuro.2016.07.005. Epub 2016 Aug 10. English, Spanish. PMID 27521134
- [Result] Zou ZJ, Liu ZH, Tang LY, Lu YP. Is there a role for extracorporeal shock wave therapy for erectile dysfunction unresponsive to phosphodiesterase type 5 inhibitors? World J Urol. 2017 Jan;35(1):167-171. doi: 10.1007/s00345-016-1899-y. Epub 2016 Jul 22. No abstract available. PMID 27447990
- [Result] Lu Z, Lin G, Reed-Maldonado A, Wang C, Lee YC, Lue TF. Low-intensity Extracorporeal Shock Wave Treatment Improves Erectile Function: A Systematic Review and Meta-analysis. Eur Urol. 2017 Feb;71(2):223-233. doi: 10.1016/j.eururo.2016.05.050. Epub 2016 Jun 16. PMID 27321373
- [Result] Kitrey ND, Gruenwald I, Appel B, Shechter A, Massarwa O, Vardi Y. Penile Low Intensity Shock Wave Treatment is Able to Shift PDE5i Nonresponders to Responders: A Double-Blind, Sham Controlled Study. J Urol. 2016 May;195(5):1550-1555. doi: 10.1016/j.juro.2015.12.049. Epub 2015 Dec 13. PMID 26694904